CLINICAL TRIAL: NCT05561036
Title: A Randomized, Double-blind, Phase Ⅲ Study of Liposomal Doxorubicin in Desmoid Tumor
Brief Title: A Randomized, Double-blind,Phase Ⅲ Study of Liposome Doxorubicin in Desmoid Tumor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Wang,MD, Chief Physician Professor, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: B2020-067-01
Record Dates: First submitted 2021-01-05; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Desmoid Tumor
Keywords: liposome doxorubicin; Desmoid Tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposome doxorubicin (Experimental): Liposome doxorubicin (50mg/m2) with a treatment cycle of once every 28 days
  Interventions: Drug: Liposome doxorubicin
- intravenous placebo (Placebo Comparator): saline solution
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Liposome doxorubicin — Liposome doxorubicin (50mg/m2) or intravenous placebo with a treatment cycle of once every 28 days
  Other Names: liposome adriamycin
  Arms: Liposome doxorubicin
Drug: Saline Solution — saline solution
  Arms: intravenous placebo

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of liposomal doxorubicin in the treatment of desmoid tumors. Unless the subject withdraws from the trial voluntarily, or the researcher considers that the subject is not suitable for further trial, each subject will be treated until the disease progresses or the toxic and side effects caused by the drug are intolerable, and then enter the survival follow-up period

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study designed to compare (PFS) differences in progression-free survival in patients treated with liposome doxorubicin or placebo. PFS is defined as the time from randomization to the first occurrence of disease progression or death caused by any cause. If the disease is stable, PFS will be calculated at the time of the last follow-up in the study. Patients who have reached the maximum follow-up period and have no progress will be reviewed on the date of the last disease assessment. The crossover data of the patients were analyzed and summarized separately from the data of the main treatment process.In this study, 72 patients were expected to be enrolled in the group for 12 months and followed up for 24 months.Patients will be randomized to receive liposome adriamycin (50mg/m2) or intravenous placebo for a treatment cycle of once every 28 days.Duration of medication: a total of 6 cycles, or to the progression of the disease, tolerable toxicity, whichever occurs first.As the disease progresses, patients treated with placebo will be allowed to enter the unblinded liposome adriamycin group.

ELIGIBILITY:
Inclusion Criteria:

* Must be confirmed as desmoid tumor by histopathology
* Patients should have measurable lesions defined by RECIST v1.1
* One of the following conditions is satisfied

  1. The disease should be defined as non resectable or tumor with disability after resection. The definition standard should meet one or more of the following characteristics

     * Multiple lesions

       * The disease has involved or does not have enough blood vessel nerve bundle, bone, skin and fascia resection boundary

         * Large tumor or multiple chambers involved
  2. Imaging showed progress (increased by 10% according to RECIST v1.1 standard size within 6 months before enrollment)
  3. The BPI score of patients with symptomatic diseases was more than 3 points and met one of the following conditions:

     * NSAIDs can not control pain, and consider increasing the control of narcotic drugs

       * Current use of narcotic drugs increased by 30%

         * New opioid anesthetics needed
* Patients are allowed to receive chemotherapy, biological (antibody) therapy, immuno or experimental therapy, tyrosine kinase inhibitors, hormone therapy or NSAIDs treatment, provided that the treatment is completed at least 4 weeks before enrollment (6 weeks of mitomycin and nitrosourea treatment) and recovers from any treatment-related toxicity below CTCAE Level 2
* Age ≥ 1 year old, male or female
* ECoG score ≤ 2
* Results of laboratory examination during screening: blood routine test: white blood cell count ≥ 3.0x 109 / L, absolute value of neutrophil ≥ 1.5 x 109 / L, platelet count ≥ 100 x 109 / L, hemoglobin ≥ 90 g / L; liver function: total bilirubin Results: serum creatinine ≤ 1.5 times of the upper limit of normal value; patients without liver metastasis had alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times of the upper limit of normal value; patients with liver metastasis had ALT and AST ≤ 5 times of the upper limit of normal value; renal function: serum creatinine ≤ 1.5 times of the upper normal value or creatinine clearance rate ≥ 50 ml / min, and urine protein < 2+
* Female subjects of childbearing age, male subjects and partners of male subjects agreed to use reliable contraceptive measures (such as abstinence, sterilization, contraceptives, contraceptive injection or subcutaneous implantation) during the study and within 6 months after the infusion of study drug)
* Understand and accept the requirements of the study, provide written informed consent and authorization for the use and disclosure of protected information, and agree to comply with the research requirements and return to conduct the required visits

Exclusion Criteria:

* Pregnant and lactating women, or fertile women who are not willing to take effective contraceptive measures during the study period
* Those who are known to be allergic to liposome doxorubicin or any component of doxorubicin, or have a history of allergy or hypersensitivity to any therapeutic component or structural analogue in this study
* Subjects previously treated with liposomal doxorubicin
* Patients who have used doxorubicin or epirubicin for more than 450 mg / m2 or more than 550 mg / m2 for epirubicin or anthracycline for heart disease
* The subjects did not receive any other drugs or anti-cancer therapy in the study
* It needs to be combined with other anti-tumor drugs
* Combined with diseases that may affect the subject's condition or ability to conduct the test, or reduce compliance, including but not limited to the following diseases:

A:Patients with active gastrointestinal bleeding, such as active peptic ulcer, ulcerative enteritis, or Crohn's disease B:Severe cardiac history: congestive heart failure > NYHA grade II; active coronary heart disease (CAD) (myocardial infarction or unstable angina pectoris, cerebrovascular disease patients within 6 months before the start of the study; uncontrolled hypertension (systolic blood pressure greater than 150 mmHg and / or diastolic blood pressure greater than 100 after combination of two or more antihypertensive drugs) MmHg) and history of hypertensive crisis or hypertensive encephalopathy C:Severe liver and kidney disease, serum ast, ALT more than 2 times the upper limit of the normal range, or Cr more than the upper limit of the normal range, total bilirubin > 1.5 times the upper limit of the normal value, patients with liver metastasis, AST and ALT > 5.0 times the upper limit of normal value D:Serious endocrine diseases, uncontrolled diabetes, blood disease, neuropsychiatric disease patients E:Patients with severe immunosuppression or long-term use of corticosteroids or immunosuppressants are known F:Active hemoptysis G:Symptomatic bacterial, fungal or viral infections, including but not limited to HIV, syphilis, or HBV or HCV infection

* Patients who have used other test drugs or devices or participated in other clinical trials within 3 months before the start of this trial
* Patients who were considered unsuitable for the trial due to other reasons

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  Progression Free Survival Rate

SECONDARY OUTCOMES:
ORR | 24 months
  Overall Response Rate
Patient Reported Outcomes-Common Terminology Criteria in Adverse Events version 5.0 | 24 months
  Patient Reported Outcomes-Common Terminology Criteria in Adverse Events version 5.0 was used to evaluate the toxicity. The evaluation time is 2 years. The data of patients who crossover or receive surgical or radiotherapy intervention will be summarized independently of their main research and treatment processes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP